CLINICAL TRIAL: NCT03867539
Title: Exparel and Education to Avoid Opioids After Carpal Tunnel Release
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kettering Health Network (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6012435
Record Dates: First submitted 2019-01-30; First posted 2019-03-08 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: hand; exparel; opioid crisis
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group; Bupivacaine + opioids (Active Comparator): This is the "standard of care" arm. This group will receive pre-operative opioid education and "standard of care", which consists of an injection of 10cc bupivacaine (plus ~1cc epinephrine and bicarbonate) into the carpal tunnel and overlying skin pre-operatively, and a post operative prescription for opioids (oxycodone/acetaminophen 5/325). Pain scores and medication usage will be tracked for three days post operatively to assess the validity and efficacy of differing pain management strategies.
  Interventions: Other: Differing pain management strategy
- Experimental Group: Exparel, no opioids (Experimental): This group will receive pre-operative opioid education, Exparel injection (liposomal bupivacaine, with bupivacaine, epinephrine and bicarbonate), and would not receive a prescription for opioids. This injection will be administered as 10cc injected in the operative field, consisting of ~5cc of Exparel (liposomal bupivacaine), ~5cc of bupivacaine, and ~1cc epinephrine. Pain scores and medication usage will be tracked for three days post operatively to assess the validity and efficacy of differing pain management strategies.
  Interventions: Other: Differing pain management strategy

INTERVENTIONS:
Other: Differing pain management strategy — The investigators aim to investigate an alternative (vs "standard") pain management strategy for post operative carpal tunnel release. All drugs used are FDA approved for these indications, and no drug itself is being investigated.

SUMMARY:
This trial seeks to use the long acting local anesthetic Exparel, in conjunction with opioid education, to attempt to avoid any post-operative opioid use following carpal tunnel surgery. This group will be compared with a "standard" group that receives non-liposomal bupivacaine, opioid education, and opioids.

DETAILED DESCRIPTION:
As has become apparent in the media, as well as in the clinical practice of nearly every type of medicine over the last few years, the nation is currently experiencing an opioid epidemic. This is a significant public health issue that has sweeping consequences that reach far beyond the medical field. The investigators believe over the last several decades, public perception regarding pain, especially post-operatively, has changed for the worse. The nation is in need of a paradigm shift in the way pain is managed, and the way the public perceives this issue, especially regarding pain expectations. As patients have become more involved with medical care as well as more knowledgeable, the investigators often see patients having performed online research regarding outcomes and expectations following particular procedures, to include post-operative pain. Commonly, even for smaller procedures performed in office, patients request opioids. As of yet, there are few data regarding use of long acting (Exparel) local analgesia alone in hand surgery, and none combining this strategy with pre-operative opioid education. The goal is to build the groundwork for the cessation of opioid prescription following carpal tunnel surgery, and produce proof that may be given patients to showing this to be an effective strategy. As some sources estimate 400,000 carpal tunnel surgeries are performed yearly, it is believed that this alternative pain management strategy, if adopted at a national level, would make a significant step towards remedying the current crisis. The rationale as to why this will be successful is the duration of action of Exparel, which has been shown to be effective for up to 72 hours. By 72 hours, post-procedure pain levels tend to have dropped precipitously, if not resolved. Use of pre-operative opioid education has also been shown to decrease perception of the need for and use of opioids. The investigators plan to study two groups: a control/standard of care group, that are given pre-operative opioid education as well as opioids, and a study group, which will have pre-operative opioid education, Exparel injection, and no opioids. Exparel will be administered as 10cc injected in the operative field, consisting of ~5cc of Exparel, ~5cc of bupivacaine, and epinephrine. All injections will be performed in the same manner. Following injection, carpal tunnel release will be performed in a similar manner in all patients. Patients that meet all of the inclusion and none of the exclusion criteria would be eligible for participation. If a patient agreed to participate, they would be randomized to group A (standard of care + education), or group B (Exparel + education + no opioids). This would be accomplished by drawing an A or B written on a paper ticket out of a bag. Adverse reactions and pain levels at 24, 48, and 72 hours will be assessed with telephone or email questionnaire, as will use of medication in the opioid group. Statistical analysis will be performed using analysis of variance, Mann-Whitney U test, and/or chi square test, as appropriate. The public health relevance of this project is to alter patient's perceived need for opioid medications post procedure, and decrease the amount of circulating opioids locally and nationally. The investigators believe this a meritorious goal, given that opioid related overdose deaths have increased eight-fold from 2012 to 2016.

ELIGIBILITY:
Inclusion Criteria:

* carpal tunnel syndrome diagnosed either by physical exam or EMG
* age >18.

Exclusion Criteria:

* allergy to bupivacaine
* pre-operative opioid usage within the last six months
* patients allergic to Percocet or acetaminophen
* patients taking tricyclic antidepressants (interaction with bupivacaine)
* vulnerable populations (prisoners or pregnant women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of post operative pain levels via Visual Analog Scale | Within the first few months of study duration
  The investigators aim to evaluate pain in either arm of the study, followed over a three day course. As several studies have shown pain to be wholly or mostly resolved by post-operative day three. Patients will answer questionnaire to include Visual Analog Scale for pain, and amount of pain medication taken. The Visual Analog Scale for pain ranges from a score of 0 to 10, with 0 being "no pain", 5 being "distressing pain", and 10 being "the worst pain imaginable"

SECONDARY OUTCOMES:
Failure of alternate pain management strategy | Within the first few months of study duration
  The investigators aim to identify any subset of patients that do not respond to combination therapy (education + Exparel). Analysis of data provided by patient-answered Visual Analog Scale will occur. Failures will be presented as a whole number and as percentage of total participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Buczek, DO, Principal Investigator — Kettering Health Network
Locations (1):
- Orthopedic Associates of Southwest Ohio, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Youha S, Lalonde DH. Update/Review: changing of use of local anesthesia in the hand. Plast Reconstr Surg Glob Open. 2014 Jun 6;2(5):e150. doi: 10.1097/GOX.0000000000000095. eCollection 2014 May. PMID 25289343
- [Background] Okamura A, Meirelles LM, Fernandes CH, Raduan Neto J, Dos Santos JB, Faloppa F. Evaluation of patients with carpal tunnel syndrome treated by endoscopic technique. Acta Ortop Bras. 2014;22(1):29-33. doi: 10.1590/S1413-78522014000100005. PMID 24644417
- [Result] Alter TH, Ilyas AM. A Prospective Randomized Study Analyzing Preoperative Opioid Counseling in Pain Management After Carpal Tunnel Release Surgery. J Hand Surg Am. 2017 Oct;42(10):810-815. doi: 10.1016/j.jhsa.2017.07.003. Epub 2017 Sep 8. PMID 28890331
- [Result] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Result] Ketonis C, Ilyas AM, Liss F. Pain management strategies in hand surgery. Orthop Clin North Am. 2015 Jul;46(3):399-408, xi. doi: 10.1016/j.ocl.2015.02.008. Epub 2015 Mar 31. PMID 26043053
- [Result] Ketonis C, Kim N, Liss F, Zmistowski B, Matzon J, Leinberry C, Wang M, Jones C, Abboudi J, Kirkpatrick W, Ilyas AM. Wide Awake Trigger Finger Release Surgery: Prospective Comparison of Lidocaine, Marcaine, and Exparel. Hand (N Y). 2016 Jun;11(2):177-83. doi: 10.1177/1558944715627618. Epub 2016 Mar 8. PMID 27390559
- [Result] Svensson I, Sjostrom B, Haljamae H. Assessment of pain experiences after elective surgery. J Pain Symptom Manage. 2000 Sep;20(3):193-201. doi: 10.1016/s0885-3924(00)00174-3. PMID 11018337